CLINICAL TRIAL: NCT02232854
Title: Comprehensive Technology-Assisted Training and Supervision Program to Enhance Depression Management in Primary Care
Brief Title: Training and Supervision Program for Depression Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Graciela Rojas Castillo, Dr.med. Psychyatrist, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1130230
Record Dates: First submitted 2014-08-07; First posted 2014-09-05 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depression training/supervision program (Experimental): A complex intervention, which will include:
  * Primary Health Care team training in depression
  * A focus group, after training
  * Telephone monitoring of patients
  * Web-based supervision of clinicians
  Interventions: Behavioral: Depression training/supervision program
- Usual Care (No Intervention): Patients in the control group will receive all the interventions that are guaranteed for persons with depression in Chile: treatment in Primary Health Care clinics with the Primary Health Care team and referral to the regional specialized psychiatric service.

INTERVENTIONS:
Behavioral: Depression training/supervision program — The intervention will be composed of:
  * Training of Primary Health Care teams to ensure compliance to the "Clinical Guidelines of the Ministry of Health for the Treatment of Depression". Primary Health Care teams will undergo an Objective Structured Clinical Examination (OSCE) for evaluation.
  * After the training, a focus group between Primary Health Care teams and study researchers will be held in order to address barriers to clinical guidelines implementation.
  * Primary Health Care clinics' trained administrative staff will contact patients from a call-center to support treatment adherence.
  * Psychiatrists, using a web-based platform, will supervise the course of the program, the allocated treatments, the patients' progress, and their response to treatment.
  Arms: Depression training/supervision program

SUMMARY:
According to the literature the management of depressive disorders at primary care level is not always consistent with guidelines. The main objective of this study is to test whether a Comprehensive Technology-Assisted Training and Supervision Program will improve depression management in Primary Health Care clinics in Santiago, Chile.

DETAILED DESCRIPTION:
A cluster randomized controlled clinical trial will be conducted in four Primary Health Care (PHC) clinics in Santiago, Chile.

The sample selection of the PHC clinics will be performed in two steps. Firstly, two urban municipalities of Santiago Metropolitan Region, Chile, will be randomly selected if they work with the Faculty of Medicine of the U.Chile and have at least two PHC.Municipalities with a high Human Development Index, high percentage of immigrants and older population, and Psychiatry residents working in PHC , will be excluded.Secondly in each selected municipalities,two PHC will be randomly selected for the active and control arm.

To detect a difference of 20%, in a one-sided model, with an alpha of 5% and power of 80%, 152 depressed persons, 76 to each group, will be required for the study. A design effect of 2.42 was estimated. After applying the design effect the sample needed increased to 368 depressed persons. Considering a retention rate of approximately 85%, 434 depressed cases will be needed required for the study, hence 109 cases in each of the 4 primary health care clinics.

Analysis and presentation of the results will be in accordance with CONSORT guidelines for randomized clinical trials, with the primary comparative analysis being conducted on an intention to treat basis and due emphasis placed on confidence intervals for the between-arm comparisons.

Initially descriptive analysis to assess the balance between two groups will be conducted. The primary analysis will employ multilevel multivariable lineal regression to investigate differences in the PHQ-9 scores between groups at 3 and 6 months after randomization, adjusting for baseline outcome variable scores. Sensitivity analysis making different assumptions will be conducted to investigate the potential effects of missing data. Similar analysis will be done for the secondary outcomes measures.

ELIGIBILITY:
Inclusion Criteria:

* signing written informed consent
* age between 18-65 years
* current depressive episode, according to the Mini-International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

* current depression treatment
* no access to telephone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Depressive Symptomatology at 3 months | Baseline , 3 months
  Depressive symptomatology measured with the Patient Health Questionnaire - Nine Item (PHQ-9) at 3 months after patient recruitment.
Change from Baseline Depressive Symptomatology at 6 months | Baseline, 6 months.
  Depressive symptomatology measured with the Patient Health Questionnaire - Nine Item (PHQ-9) at 6 months after patient recruitment.

SECONDARY OUTCOMES:
Adherence to depression treatment at patient's level | 3 and 6 months after baseline.
Change from Baseline Quality of life at 3 and 6 months | Baseline , 3 months, 6 months.
  Quality of life at patient's level measured with the Health Survey, Short form (SF-36), at 3 months and 6 months after patient recruitment.
Change from Baseline Clinical Outcomes at 3 and 6 months | Baseline , 3 months, 6 months.
  Clinical outcomes at patient's level measured with the Outcome Questionnaire-45.2 (OQ-45.2), at 3 months and 6 months after patient recruitment.
Use of Health Care services at patient's level | 3 and 6 months after baseline
  Use of Health Care services at patient's level measured with and ad-hoc built questionnaire.
Rate of treated depressed cases at Primary Care team level | 12 months before randomization and 12 months after.

CONTACTS AND LOCATIONS:
Locations (4):
- Chile (4):
  - CESFAM Garín, Quinta Normal, Santiago Metropolitan
  - CESFAM Lo Franco, Quinta Normal, Santiago Metropolitan
  - CESFAM Barros Luco, San Miguel, Santiago Metropolitan
  - CESFAM Recreo, San Miguel, Santiago Metropolitan

REFERENCES:
- [Derived] Rojas G, Martinez P, Vohringer PA, Martinez V, Castro-Lara A, Fritsch R. Comprehensive technology-assisted training and supervision program to enhance depression management in primary care in Santiago, Chile: study protocol for a cluster randomized controlled trial. Trials. 2015 Jul 24;16:311. doi: 10.1186/s13063-015-0845-4. PMID 26201546